CLINICAL TRIAL: NCT06722911
Title: Nimotuzumab Combined with Nab-paclitaxel+ Gemcitabine As Postoperative Adjuvant Therapy in Patients with EGFR-positive Pancreatic Cancer: a Prospective, Single-arm Study
Brief Title: Study of Adjuvant Nimotuzumab Combined with Nab-paclitaxel+ Gemcitabine in EGFR-positive Pancreatic Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IST-Nim-PC-42
Record Dates: First submitted 2024-12-04; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Pancreatic Cancer Resectable
MeSH Terms: interventions — nimotuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nimotuzumab+ AG (Experimental)
  Interventions: Drug: Nimotuzumab; Drug: AG

INTERVENTIONS:
Drug: Nimotuzumab — Nimotuzumab 400 mg on Day 1 and 15 of a 28-day cycle (6 cycles) ; Patients will receive Nimotuzumab 600 mg on days 1 and 8 of every 21-day cycle. Patients will receive six treatment cycles unless there is radiologic evidence of disease recurrence and unacceptable toxicity.
Drug: AG — Patients will receive nab-paclitaxel 125 mg/m^2 followed by gemcitabine 1,000 mg/m^2 as one intravenous infusion over 30-40 minutes on days 1 and 8 of every 21-day cycle. Patients will receive six treatment cycles unless there is radiologic evidence of disease recurrence and unacceptable toxicity.

SUMMARY:
This is a prospective, single-arm trial. The main purpose of the study is to evaluate the efficacy and safety of Nimotuzumab combined with nab-paclitaxel+ gemcitabine (AG regimen) for postoperative adjuvant treatment of pancreatic cancer with EGFR-positive.

DETAILED DESCRIPTION:
This clinical study is designed as a prospective, open-label, single arm, phase II study to evaluate the clinical efficacy and safety of Nimotuzumab combined with AG (nab-paclitaxel+ gemcitabine) as postoperative adjuvant therapy in patients with EGFR-positive pancreatic cancer. The main endpoint is disease-free survival (DFS). Additional end points included distant metastasis-free survival (DMFS), overall survival (OS), tumor-related markers and safety.

ELIGIBILITY:
Inclusion Criteria:

* 1. Able and willing to provide a written informed consent.
* 2. Age 18-75 years old, gender unlimited;
* 3. Histologically or cytologically confirmed resected pancreatic ductal adenocarcinoma (PDAC), resectable evaluation is based on criteria of NCCN guidelines, no evidence of distant metastasis as demonstrated by imaging;
* 4. Postoperative pathology suggested R0/R1 resection;
* 5. EGFR positive (by immunohistochemistry);
* 6. KRAS gene and CDX-2 protein status must have been determined at baseline (only for post hoc analysis);
* 7. Adequate organ and bone marrow function, defined as follows: absolute neutrophil count (ANC)≥1.5×10^9/L; platelets≥80×10^9/L; hemoglobin≥9.0 g/dL; serum total bilirubin (TBIL)≤1.5×ULN; aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 times the upper limit of normal (ULN); serum creatinine≤1.5×ULN or estimated creatinine clearance > 60 mL/min;
* 8. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
* 9. Postoperative survival is expected to be ≥3 months;
* 10. Fertile subjects are willing to take contraceptive measures during the study period.

Exclusion Criteria:

* 1. Prior neo-adjuvant treatment, radiation therapy, or systemic therapy for pancreatic adenocarcinoma;
* 2. History of other malignancies (except cured basal cell carcinoma of the skin and carcinoma in situ of the cervix);
* 3. Accompanied by other serious diseases, including but not limited to: compensatory heart failure (NYHA grade III and IV), unstable angina, poorly controlled arrhythmias, uncontrolled hypertension (SBP>160mmHg or DBP>100mmHg); active infections; unmanageable diabetes mellitus; presence of uncontrolled pleural effusion, pericardial effusion, or ascites requiring drainage; severe portal hypertension; gastric outlet obstruction; Respiratory insufficiency;
* 4. Postoperative complications such as bleeding, pancreatic fistula, gastric obstruction, abdominal infection, and biliary fistula, which made the patient unable to receive adjuvant therapy within 12 weeks after surgery;
* 5. CA199>180 U/ml within 21d before adjuvant therapy;
* 6. Known allergy to prescription or any component of the prescription used in this study;
* 7. Known HIV, or syphilis infection, or active hepatitis (hepatitis B, hepatitis C);
* 8 .Other reasons that are not suitable to participate in this study according to the researcher's judgment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
disease-free survival (DFS) | Up to 24 months
  The time from the date of surgery to the disease recurrence or death, whichever is earlier.

SECONDARY OUTCOMES:
distant metastasis-free survival (DMFS) | Up to 24 months
  The time from the date of surgery to the first distant metastasis or death due to any cause, whichever is earlier.
overall survival (OS) | Up to 24 months
  The time from the date of surgery to death due to any cause.
tumor-related markers | Up to 24 months
  To explore the influence of tumor-related markers (such as KRAS gene, CDX-2 protein, etc.) on prognosis.
adverse events | Up to 30 days after last administration
  Frequency and severity of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Yiping Mou, Dr, Study Chair — Zhejiang Provincial People's Hospital
Locations (1):
- Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No